CLINICAL TRIAL: NCT04263740
Title: The Efficacy of Kinesio Taping as an Adjunct Intervention to Traditional Physical Therapy in the Treatment of Nonspecific Acute Low Back Pain: A Prospective Randomized Controlled Trial
Brief Title: The Efficacy of Kinesio Taping in the Treatment of Nonspecific Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rocky Mountain University of Health Professions (Other)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Prof. Dr Mahmoud Ibrahim Ibrahim, Professor of orthopedic PT, Rocky Mountain University of Health Professions
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05291519Exp
Record Dates: First submitted 2020-02-04; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: This study followed a prospective experimental pretest-posttest control group randomized design with repeated measures. Two groups were included in this study, an experimental group and a control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding the physical therapist (the principal investigator) who provided interventions to both groups in the study to the type of intervention was not feasible. Blinding the principal investigator to the assessment process was possible by using another physical therapist who conducted all measurements. Blinding the assessor to subject's group assignment was done to ensure unbiased ascertainment of outcomes. Randomization also served to reduce the risk of selection bias by the principal investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping plus Traditional Physical Therapy (Experimental): Kinesio Taping plus Traditional physical therapy
  Interventions: Procedure: Kinesio Taping; Procedure: Traditional Physical therapy
- Traditional Physical Therapy (Other): Traditional physical therapy was in the form of patient education, manual therapy and therapeutic exercises.
  Interventions: Procedure: Traditional Physical therapy

INTERVENTIONS:
Procedure: Kinesio Taping — Taping for 3 days every week and two sessions of PT twice a week. The PI also instructed the patient to inform him if the tape gets off or become loose. KT was removed after 72 hours, and then reapplied after a few days rest to allow the skin to recover and to avoid skin irritation. The patient was instructed to refrain from getting the tape wet for 30 to 45 minutes after application to allow for better adherence. Patients were also instructed to be careful during dressing and undressing so the tape does not get caught with their clothes if the edges of the tape get slightly loose. No physical therapy treatment or taping was provided during the rest period except for the prescribed home exercise program. Patients in both groups received the same traditional physical therapy treatment two times a week.
  Arms: Kinesio Taping plus Traditional Physical Therapy
Procedure: Traditional Physical therapy — Traditional physical therapy was in the form of patient education, manual therapy and therapeutic exercises. Patient education focused on the natural history of the condition and its favorable prognosis, positive thinking, and encouragement of activity participation. Patient education was delivered through one-on-one discussion by the principal investigator.

SUMMARY:
The Purpose of the study was to examine the effect of KinesioTaping (KT) on disability, fear avoidance beliefs and pain intensity in patients with acute non-specific LBP. Materials and Methods: Seventy-eight patients were randomized to an experimental group that received traditional physical therapy plus KT and a control group that received traditional physical therapy alone. Interventions were administered twice a week for four weeks. Assessment tools used were; RMDQ for disability, FABQ for fear-avoidance beliefs and NPRS for pain intensity.

DETAILED DESCRIPTION:
This study followed a prospective experimental pretest-posttest control group randomized design with repeated measures. Two groups were included in this study, an experimental group and a control group. Both groups were tested with respect to three main outcomes which are disability, fear avoidance beliefs and pain intensity. Five points of measurements were used; at baseline, at the end of week 1, at the end of week 2, at the end of week 3 and at the end of week 4.

A total of 88 patients with a primary complaint of low back pain were enrolled and consented to participate in the study. Potential study participants were assessed for study eligibility based on the pre-defined inclusion and exclusion criteria. Study flow chart. Subjects were pre-screened for known contraindications and precautions to thrust joint manipulation and exercises. No individuals were excluded from participation in this study based on race, creed, color, gender, age, national or ethnic origin, sexual orientation, disability, or health status.

After obtaining the informed consent, participant's demographic information was collected including age, gender, ethnicity, contact information, emergency contact, employment status etc. History taking also included collecting information about patient's past medical history, family history, mechanism of injury, chief complaint, present history, number of days since onset, presence of previous episodes of low back pain, treatment for previous episodes, questions related to red flags, and review of systems and allergies. Patients were also checked for eligibility criteria. Pain characteristics were also documented including, pain intensity, location, duration, timing, character, aggravating and alleviating factors. History, review of systems and medical screening questionnaire were also used to identify red flags. Red flags are clinical features that may indicate a serious spinal pathology that warrant further investigation.

Each participant was examined by the PI who conducted a thorough physical exam that included observation, palpation, and assessment of vertebral mobility, range of motion testing, muscle tests, neurological screening and special tests. Neurological examination included sensation for dermatomes, muscle testing for myotomes and deep tendon reflexes (Knee jerk and Ankle jerk). The allergy test for Kinesio taping was performed for all participants by the PI. An I strip of KT was applied on either side of lumbar spine at around 25% tension and left in place for 24 hours. The patient was checked during the second visit for any signs of adverse reactions such as rash or excessive hotness or itching in the tested area.

The PI then opened a new file for the participant that included all the information obtained from history taking, physical examination and any other assessments. This process took between 30 minutes and 45 minutes. In the second visit, the tape was removed and the patient checked for any abnormal reactions. The participant was then randomized to either the experimental group or the control group using random number generator.

The PI provided the research assistant with participant's basic information including the case number but the research assistant was not aware of the participant group allocation. The research assistant then performed all baseline outcome assessments required for the study which included disability as measured with the Ronald Morris Disability Questionnaire, fear avoidance beliefs as measured with Fear Avoidance Beliefs Questionnaire and pain as measured with the Numerical Pain Rating Scale. The research assistant conducted all study related measurements at baseline (W0), at the end of the first week (W1), at the end of the second week (W2), at the end of the third week (W3) and at the end of the fourth week (W4) and kept all data in a separate locked file cabinet. The second visit took approximately between 45 and 60 minutes to be completed including providing first treatment session. Assessments of study variables took 15 to 20 minutes.

A priori analysis was conducted with an alpha level (α) of 0.05, an effect size of 0.25 and a power of 80 % using G*Power (Version 3.0.10). The results indicated that a total 78 subjects would be needed of two groups. However, considering a potential 10-15 % dropout or loss to follow-up rate, around 42 to 45 participants were considered for each group.

Blinding the physical therapist (the principal investigator) who provided interventions to both groups in the study to the type of intervention was not feasible. Blinding the principal investigator to the assessment process was possible by using another physical therapist who conducted all measurements. Blinding the assessor to subject's group assignment was done to ensure unbiased ascertainment of outcomes. Randomization also served to reduce the risk of selection bias by the principal investigator. An online random number generator available at http://www.graphpad.com/quickcalcs/randomize1/ was used to randomly assign participants to two equal groups. The study was conducted at Quick Docs Medical Center located in Brooklyn, NY. This facility is the primary place of employment of the principal investigator and the research assistant. The facility has private treatment rooms where each subject was interviewed and assessment and intervention sessions were conducted. All research activities were approved by the IRB of NOVA Southeastern University. IRB approval was granted on the 29th of June of 2015. All patients provided informed consent prior to participation.

The outcome variables which were included in the study are; disability, fear-avoidance beliefs and pain intensity. The primary outcome was disability and the secondary outcomes were fear avoidance beliefs and pain intensity. Disability was evaluated with the Ronald-Morris Disability Questionnaire (RMDQ). RMDQ is a patient reported outcome measure that is composed of 24 yes/no questions to assess functional status and disability in patients with low back pain. RMDQ scores can range from 0, the highest functional status indicating no disability, to 24, the lowest functional status indicating maximum disability. Patients were asked to mark the sentences that describe them at the time of evaluation.

Fear avoidance beliefs questionnaire (FABQ) is an assessment tool that is developed based on the fear avoidance model of exaggerated pain perception. This model is a theoretical approach of analyzing the behavior of patients with acute conditions as some of these patients recover successfully while others develop chronic pain. FABQ measures patient's fear of pain in terms of patients' behavior as a result of pain in relation to general physical activities and work related functions because of their fear. It consists of two subscales, a work subscale and a physical activity subscale; each item is scored from 0 to 6. Greater fear and consequent avoidance beliefs are associated with higher scores.

Assessment of pain was done using the numerical rating of pain scale (NPRS), which is an 11-point scale from 0 to 10, 0 indicating "no pain" and 10 indicating "the worst pain". Pain assessments were conducted at baseline and at the end of each week, for four weeks. A verbal response was required from each participant. Three measurements were taken, the current pain level, the worst pain level over the last 24 hours and the lowest pain level over the last 24 hours. The average of the three readings was used as the average pain level for each participant.

Descriptive statistics was conducted to describe all basic characteristics of participants of both groups. Variables such as age, gender, presence of previous episodes, and duration of the current episode were described. Graphical representation of the above-mentioned variables as well as the main outcome measures were obtained from statistical software. Tables and figures were used to provide an understanding of all relevant study data. Mixed model analysis of variance (ANOVA) was used to reveal main effects and interaction effects. The group type was the between-subjects' variable and the time was the within subjects' variable. Bonferroni post-tests were used to compare between groups at each individual point of time. SPSS Version 23.0 (SPSS, Inc., IBM Corporation, Somers, New York) and GraphPad Prism (Version 6.01 for Windows; GraphPad Software, San Diego, CA, USA) were used for statistical analysis.

All patients' data and records pertaining to this research study and any relevant information were stored in a locked file cabinet at the facility in which the study was conducted. A case number was used to indicate patient's identity on these records. This information was only accessible to the principal investigator, the independent physical therapist, and other research study staff involved in conducting this research study. All assessment data were kept in a separate locked file cabinet which was accessible only to the independent physical therapist. To ensure confidentiality, no confidential information such as patient's name, address, phone number, or any other information that might possibly be used to link the data to the patient was transmitted or shared. These measures were used to ensure patients' confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, age between 18 and 75.
* Primary complaint of pain in the lower back located between the costal margins and the gluteal folds, less than 4 weeks in duration with or without leg pain but symptoms not distal to the knee.
* A new episode of low back pain. This is defined as an episode which was preceded by a period of at least one month without low back pain where the participant was not consulting a health care practitioner or taking medication for their low back pain.
* Pain of sufficient intensity to interfere with patient's daily activities and function. A minimum pain intensity of 3 on the numerical pain rating scale to allow room for change, as the MCID for the NPRS is 2 points. A minimal score of 4 on the RMDQ will also be required as patients with scores under 4 and over 20 may not show meaningful change over time. NPRS and RMDQ were used to determine such criteria.
* Ability to communicate with English language which is important to complete the questionnaires successfully.
* Lumbar spine hypomobility. This was determined through palpation by applying postero-anterior pressure by the tips of the thumbs against the spinous processes of all segments of the lumbar spine. Three oscillatory postero-anterior movements were performed at each level. Through comparison of quality and range of movements at each level, the physical therapist can determine which segments are stiff or hypomobile and the quality of the end feel.

Exclusion Criteria:

* Patients with a diagnosis of severe degenerative and stenotic conditions which make spinal manipulative therapy contraindicated.
* known or suspected serious spinal pathology (metastatic tumors, inflammatory or infective diseases of the spine, cauda equina syndrome, spinal fracture, dislocations/sublaxations).
* Nerve root compromise evidenced by at least two of the following (a) myotomal weakness, (b) dermatomal or widespread sensory loss, (c) hypo or hyper-reflexia of the lower limb reflexes. Examination of sensation, reflexes and motor power were used to identify such criteria.
* Adverse skin reactions to Kinesio taping.
* RMDQ score of less than 4 or more than 20.
* NPRS of less than 3.
* Patients taking NSAIDs.
* Patients currently receiving physical therapy or any form of manual therapy.
* Previous spinal surgery.
* Patients with contraindications to manual therapy or therapeutic exercises.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2016-04-28 (Actual)

PRIMARY OUTCOMES:
Disability | changes at five points of time, at baseline (W0, before interventions), at the end of the first week (W1), at the end of the second week (W2), at the end of the third week (W3) and at the end of the fourth week (W4).
  Disability was evaluated with the Ronald-Morris Disability Questionnaire (RMDQ). RMDQ is a patient reported outcome measure that is composed of 24 yes/no questions to assess functional status and disability in patients with low back pain. RMDQ scores can range from 0, the highest functional status indicating no disability, to 24, the lowest functional status indicating maximum disability. Patients were asked to mark the sentences that describe them at the time of evaluation.

SECONDARY OUTCOMES:
Fear avoidance beliefs questionnaire (FABQ) | changes at five points of time, at baseline (W0, before interventions), at the end of the first week (W1), at the end of the second week (W2), at the end of the third week (W3) and at the end of the fourth week (W4).
  Fear avoidance beliefs questionnaire (FABQ) is an assessment tool that is developed based on the fear avoidance model of exaggerated pain perception.36-38 This model is a theoretical approach of analyzing the behavior of patients with acute conditions as some of these patients recover successfully while others develop chronic pain.37,38 FABQ measures patient's fear of pain in terms of patients' behavior as a result of pain in relation to general physical activities and work related functions because of their fear. 37,38 It consists of two subscales, a work subscale and a physical activity subscale; each item is scored from 0 to 6. Greater fear and consequent avoidance beliefs are associated with higher scores.
Assessment of Pain | changes at five points of time, at baseline (W0, before interventions), at the end of the first week (W1), at the end of the second week (W2), at the end of the third week (W3) and at the end of the fourth week (W4).
  Assessment of pain was done using the numerical rating of pain scale (NPRS), which is an 11-point scale from 0 to 10, 0 indicating "no pain" and 10 indicating "the worst pain".39 Pain assessments were conducted at baseline and at the end of each week, for four weeks. A verbal response was required from each participant. Three measurements were taken, the current pain level, the worst pain level over the last 24 hours and the lowest pain level over the last 24 hours. The average of the three readings was used as the average pain level for each participant.

IPD SHARING:
Plan to Share IPD: Yes
we can share raw data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: upon approval for 10 years
Access Criteria: only for meta analysis and additional research

DOCUMENTS (1):
  • Informed Consent Form (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT04263740/ICF_000.pdf